CLINICAL TRIAL: NCT05896982
Title: Optimizing Patient Experience During Myocardial Perfusion Imaging
Acronym: OPTIMIZE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tilburg University (Other)
Collaborators: Elisabeth-TweeSteden Ziekenhuis (Other); Verbeeten Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: NL81600.028.22
Record Dates: First submitted 2023-03-15; First posted 2023-06-09 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-04

CONDITIONS: Myocardial Ischemia; Myocardial Infarction; Autonomic Dysfunction
MeSH Terms: conditions — Myocardial Ischemia; Myocardial Infarction; Primary Dysautonomias

STUDY DESIGN:
Intervention Model Description: Experimental 2x2 factorial design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Care as usual (No Intervention): Patients in this group will not receive any additional information materials or support on top of care as usual, but information videos will be made available after completion of the MPI procedures.
- Care as usual with information support (Experimental): Patients in this group will primarily receive additional information on the diagnostic process that they will go through with the use of video materials. Supportive coaching will not be provided in this group.
  Interventions: Other: Care as usual with information support
- Care as usual with supportive coaching (Experimental): Patients in this group will receive supportive coaching throughout their clinic visit. The coach is available for questions as well as specific support for each patient. Information support using video materials will not be supplied to the patients during the diagnostic process in this group, but will be made available after completion of the MPI procedures.
  Interventions: Other: Care as usual with supportive coaching
- Care as usual with information support and supportive coaching (Experimental): Patients in this group will receive both information support as well as supportive coaching during their diagnostic clinic visit.
  Interventions: Other: Care as usual with information support and supportive coaching

INTERVENTIONS:
Other: Care as usual with information support — Comprises of additional visual information in the form of two videos that show details about the procedure on both days of the MPI diagnostic procedure. Each of these two videos are approximately 5 minutes long and are made available to the patients before the first day (video 1), and in between the first and second day (video 2).
  Arms: Care as usual with information support
Other: Care as usual with supportive coaching — Patients receive coaching from one person who is present throughout the complete diagnostic process. The coach is available for answering questions as well as comforting the patients when necessary (e.g., to reassure patients if they are anxious or stressed).
  Arms: Care as usual with supportive coaching
Other: Care as usual with information support and supportive coaching — This intervention comprises additional visual information in the form of two videos and coaching throughout the diagnostic process as described above.
  Arms: Care as usual with information support and supportive coaching

SUMMARY:
The present study focusses on the effects of the diagnostic testing environment on psychological wellbeing, cardiac symptoms and patient satisfaction during cardiac stress testing (CST) in patients who are referred to the Institute Verbeeten for SPECT myocardial perfusion imaging (MPI).

The diagnostic procedure consists of two days of MPI using SPECT: day 1 of MPI involves obtaining a resting image and day 2 (typically 3 or 4 days later) a stress MPI following exercise or pharmacological challenge with adenosine. The diagnostic procedure can result in undesirable effects on psychological wellbeing, such as anxiety or psychological distress. These effects can be related to anticipatory anxiety (day 1 of MPI) and/or responses to the exercise or adenosine stress testing (day 2 of MPI). The present investigation aims to develop methods to further improve patients' experiences and wellbeing during the diagnostic process for the presence of inducible myocardial ischemia.

This research project will compare four groups to establish the effect of providing information and supportive coaching: (1) care as usual, (2) information support using video materials, (3) supportive coaching during the diagnostic testing procedure, and (4) a combination of both interventions. The video-based information and supportive coaching are aimed at reducing feelings of anxiety, uncertainty and psychological distress during the diagnostic testing procedure. In addition to standardized self-report questionnaires, this project will utilize facial expression analysis software to measure emotional states during CST as well as 24- hour ambulatory assessments to evaluate autonomic nervous system activity, cardiac symptoms and psychological wellbeing during everyday life activities in the period between the two days of MPI. It is hypothesized that additional video-based information and supportive coaching during the diagnostic process for the inducibility of myocardial ischemia will result in improved psychological wellbeing (reduced acute negative emotions; primary outcome) as well as less cardiac and other physical symptoms and improved patient satisfaction (secondary outcomes) of the diagnostic clinic visit. The innovative aspect of the present proposal is its focus on emotional expression during evaluation for myocardial ischemia using FaceReader software in combination with self-reported momentary mood and perceived stress assessments. Knowledge about the interaction between psychological wellbeing and cardiac function obtained in this project will strengthen the development of future interventions aimed to reduce symptom burden and psychological distress in patients undergoing diagnostic evaluations for heart disease.

ELIGIBILITY:
Inclusion Criteria:

* referred to the Institute Verbeeten Tilburg and eligible for adenosine-exercise SPECT MPI
* capable of answering questionnaires and receiving information and coaching in Dutch.

Exclusion Criteria:

* a life-threatening disease with < 1 year survival (e.g., metastatic cancer)
* refusal to informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Psychological wellbeing - self report using Profile of Mood States | During the two day diagnostic process.
  Will be assessed using self-report measures of emotional states on a scale from 0 to 10 (stressed, anxious, insecure, relaxed, worried, irritated, excited, and tired) with a higher score representing more of this emotional state.These measures of psychological well-being will be compared between the four groups.
Psychological wellbeing - Facial expressions of emotions | During the stress test on day 2.
  Will be assessed using facial expression of emotions based on video recordings during the diagnostic testing procedure. Facial expressions will be analyzed (valence and intensity; e.g., anxiety) using FaceReader software as in our prior METC-approved research projects at Institute Verbeeten. A value between 0 and 1 will be the outcome measure for each emotion (happy, sad, angry, surprised, scared, disgusted and neutral). These measures of psychological well-being will be compared between the four groups.

SECONDARY OUTCOMES:
Cardiac symptoms | During the two day diagnostic process.
  The intensity of cardiac symptoms and other common symptoms during MPI SPECT (e.g., headache, dizziness, fatigue, nausea) will be assessed using self-report measures on a scale from 0 to 10. Higher scores represent a higher intensity of the symptoms.
Patient experience - PSQ-18 | At the end of the two day diagnostic process.
  Patient experience and satisfaction of the clinic visit, cardiac tests, and coaching will be assessed using a validated questionnaire with a higher score representing a better patient experience.
Physiological measures - heart rate | During the cardiac stress test on the second day of the diagnostic process.
  During the cardiac stress test, heart rate is routinely collected. This data will be used as a physiological measure that is relevant to emotional experiences, cardiac symptoms, and the inducibility of myocardial ischemia.
Physiological measure - blood pressure | During the cardiac stress test on the second day of the diagnostic process.
  During the cardiac stress test, blood pressure is routinely collected. This data will be used as a physiological measure that is relevant to emotional experiences, cardiac symptoms, and the inducibility of myocardial ischemia.
Ambulatory ECG monitoring | For 24 hours between the first and second day of the diagnostic process.
  A 24-hour Holter-ECG will be used to assess heart rate variability during everyday life activities. These assessments are obtained out-of-clinic during the day between the resting and stress MPI SPECT assessment.
SPECT images | At the end of the first and second day of the diagnostic process.
  As part of the patient's clinical care, single-photon emission computed tomography will be used to obtain myocardial perfusion images on the rest and cardiac stress test days. The presence or absence of ischemia can be evaluated based on these images.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute Verbeeten, Tilburg, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adelstein SJ. Administered radionuclides in pregnancy. Teratology. 1999 Apr;59(4):236-9. doi: 10.1002/(SICI)1096-9926(199904)59:43.0.CO;2-6. PMID 10331526
- [Background] Baik SH, Fox RS, Mills SD, Roesch SC, Sadler GR, Klonoff EA, Malcarne VL. Reliability and validity of the Perceived Stress Scale-10 in Hispanic Americans with English or Spanish language preference. J Health Psychol. 2019 Apr;24(5):628-639. doi: 10.1177/1359105316684938. Epub 2017 Jan 5. PMID 28810432
- [Background] Bekendam MT, Mommersteeg PMC, Vermeltfoort IAC, Widdershoven JW, Kop WJ. Facial Emotion Expression and the Inducibility of Myocardial Ischemia During Cardiac Stress Testing: The Role of Psychological Background Factors. Psychosom Med. 2022 Jun 1;84(5):588-596. doi: 10.1097/PSY.0000000000001085. Epub 2022 Apr 14. PMID 35420591
- [Background] Bekendam MT, Vermeltfoort IAC, Kop WJ, Widdershoven JW, Mommersteeg PMC. Psychological factors of suspect coronary microvascular dysfunction in patients undergoing SPECT imaging. J Nucl Cardiol. 2022 Apr;29(2):768-778. doi: 10.1007/s12350-020-02360-5. Epub 2020 Oct 6. PMID 33025473
- [Background] Bekendam MT, Kop WJ, Vermeltfoort IAC, Widdershoven JW, Mommersteeg PMC. Facial Expressions of Emotions During Pharmacological and Exercise Stress Testing: the Role of Myocardial Ischemia and Cardiac Symptoms. Int J Behav Med. 2021 Dec;28(6):692-704. doi: 10.1007/s12529-021-09963-3. Epub 2021 Feb 23. PMID 33619698
- [Background] Bekendam MT, Mommersteeg PMC, Kop WJ, Widdershoven JW, Vermeltfoort IAC. Anxiety and hemodynamic reactivity during cardiac stress testing: The role of gender and age in myocardial ischemia. J Nucl Cardiol. 2021 Dec;28(6):2581-2592. doi: 10.1007/s12350-020-02079-3. Epub 2020 Feb 28. PMID 32112295
- [Background] Gabbay FH, Krantz DS, Kop WJ, Hedges SM, Klein J, Gottdiener JS, Rozanski A. Triggers of myocardial ischemia during daily life in patients with coronary artery disease: physical and mental activities, anger and smoking. J Am Coll Cardiol. 1996 Mar 1;27(3):585-92. doi: 10.1016/0735-1097(95)00510-2. PMID 8606268